CLINICAL TRIAL: NCT01053897
Title: A Phase 2, Multicenter, Double-Blind, Placebo-Controlled Study of GBT009 for Treatment of Incisional Wounds Following Breast Reconstruction Surgery
Brief Title: Study of GBT009 for Treatment of Incisional Wounds Following Breast Reconstruction Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Garnet BioTherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBT-09-001
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2013-10-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-08

CONDITIONS: Scar Formation
Keywords: GBT009; incisional scar; breast reconstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GBT009 (Experimental)
  Interventions: Biological: GBT009
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GBT009 — Intradermal Injection following surgery
  Arms: GBT009
Biological: Placebo — Intradermal Injection following surgery
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess whether intradermal injections of GBT009 along full thickness incisions following surgery results in an improvement in scar appearance.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following criteria to be considered eligible to participate in the study:

* be a female between 18 and 70 years of age, inclusive
* have a body mass index ≤ 32 kg/m2 and a body weight between 50 and 95 kg, inclusive
* be scheduled for a mastectomy with breast reconstruction surgery using an abdominal flap technique
* for women diagnosed with breast cancer, has standard of care treatment for breast cancer prior to surgery and will have standard of care treatment for breast cancer after surgery
* for subjects of childbearing potential, be surgically sterile or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA through completion of the study and have negative results on a serum pregnancy test done before administration of study medication (women who are postmenopausal [no menses for at least 2 years] are also eligible to participate)
* be able to understand the study procedures, agree to participate in the study program, and voluntarily provide written informed consent

Exclusion Criteria: Subjects who meet any of the following criteria will be excluded from participating in the study:

* have clinically significant laboratory abnormalities at screening
* have, as determined by the investigator or the sponsor's medical monitor, a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, coagulopathic disorder or other condition that would preclude participation in the study
* have received treatment for a severe, uncontrolled inflammatory disease or allergic condition within three months of screening
* have a life expectancy ≤ 2 years
* have a history of alcoholism or drug addiction or abuse within 5 years
* have evidence of a clinically significant abnormality upon evaluation of 12 lead ECG
* have evidence of any past or present clinically significant medical condition, including skin disease, that would impair wound healing
* have a history of keloid scar formation
* have existing scarring in the abdominal area of study that would interfere with the efficacy assessments
* have a history of (within the past 5 years) or an active malignancy, other than breast cancer
* have a breast cancer that has been staged at Stage IIIB, IIIC or IV
* have received a cytotoxic agent or have been treated with radiation within 90 days of screening and/or, in the opinion of the investigator, will likely require treatment in the 30 day period following the administration of study medication
* have received anticoagulation medication within 5 days of dosing with study medication
* have participated in any study involving an investigational product within 30 days before dosing with study medication
* have routinely used tobacco products within 6 months preceding the study period

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garnet Study Manager, Study Director — Garnet BioTherapeutics, Inc.
Locations (2):
- United States (2):
  - Garnet BioTherapeutics Investigational Site, Chicago, Illinois
  - Garnet BioTherapeutics Investigational Site, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at two US centers (surgical practices) beginning in February 2010. The last subject completed participation in October 2011
Groups:
- GBT009/Placebo: All subjects acted as their own control receiving both GBT009 and Placebo
Period: Overall Study
Arm/Group | GBT009/Placebo
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GBT009/Placebo
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Photography- Independent Scar Assessment Panel
Description: An independent panel was planned to review scar photography to determine more preferable outcomes. Panel was not performed.
Time Frame: 0.5, 1, 2, 3, 6, 9 and 12 Months
Population: All subjects had scar photography completed at study visits. However, due to the early termination of this trial, the independent panel review was not completed.
Groups:
- GBT009; Placebo: All subjects acted as their own control receiving both GBT009 and Placebo
Arm/Group | GBT009 | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Scar Preference
Description: Overall preference of the healing/appearance of each scar segment as completed by investigator and subject.
Time Frame: 12 Month (End of Study)
Population: All Subjects included.
Measure: Number; unit: participants
Groups:
- GBT009: GBT009 treated scar segment preferred
- Placebo: Placebo treated scar segment preferred
- No Difference: No scar segment was preferred to the other
Arm/Group | GBT009 | Placebo | No Difference
Number analyzed (Participants) | 5 | 5 | 5
participants
  Investigator Evaluation | 4 | 0 | 1
  Subject Evaluation | 2 | 2 | 1

3. Secondary Outcome: Patient Observer Scar Assessment Scale (POSAS)
Description: Rating by subject and investigator (observer) to assess various factors of scar segment appearance/characteristics on a numeric scale (0-10). Individual parameters rated by the subject or observer according to a 0-10 scale where 0 equals no symptoms or difference from normal (better) and 10 equals the worst possible symptoms or difference from normal (worse).
  Outcomes measured at 0.5, 1, 2, 3, 6, 9 and 12 Months. Reported Data is end of study (12 months)
Time Frame: 12 Month (End of Study)
Population: All subjects were included
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- GBT009: Therapy treated scar segment
- Placebo: Placebo treated scar segment
Arm/Group | GBT009 | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale
  Vascularization (Observer) | 4.8 (1.79) | 4.6 (1.82)
  Pigmentation (Observer) | 4.4 (1.14) | 4.4 (1.52)
  Thickness (Observer) | 3.4 (2.07) | 2.6 (1.52)
  Relief (Observer) | 3.6 (1.82) | 3.4 (1.52)
  Pliability (Observer) | 3 (1.41) | 2.4 (1.52)
  Pain (Subject) | 1 (0) | 1 (0)
  Itching (Subject) | 1 (0) | 1 (0)
  Color (Subject) | 5.4 (2.88) | 4.6 (3.20)
  Stiffness (Subject) | 3.4 (3.78) | 3 (3.94)
  Thickness (Subject) | 3.8 (3.56) | 3.8 (3.70)
  Irregularity (Subject) | 4 (2.74) | 4 (2.65)

4. Secondary Outcome: Manchester Scar Scale (MSS)
Description: Rating by investigator to assess various factors of scar appearance/characteristics on numeric scales.
  MSS includes a visual analog scale (10 cm; 0 excellent appearance, 10 poor appearance) and four descriptive characteristics rated 1 to 4 according to the following descriptions.
  Color: Perfect (1), Slight mismatch (2), Obvious mismatch (3), Gross mismatch (4).
  Contour: Flush with surrounding skin (1), Slightly proud/indented (2), Hypertrophic (3), Keloid (4).
  Distortion: None (1), Mild (2), Moderate (3), Severe (4). Texture: Normal (1), Just palpable (2), Firm (3), Hard (4).
  Outcomes measured at 0.5, 1, 2, 3, 6, 9 and 12 Months. Reported Data is end of study (12 months)
Time Frame: 12 Month (End of Study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GBT009 | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale
  Visual Analog Scale (0-10) | 4.26 (2.62) | 4.26 (2.32)
  Color (1-4) | 2.6 (0.55) | 2.4 (0.55)
  Contour (1-4) | 1.6 (0.55) | 1.4 (0.55)
  Distortion (1-4) | 1.8 (0.45) | 1.8 (0.45)
  Texture (1-4) | 4.8 (1.79) | 4.6 (1.82)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | GBT009/Placebo
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBT009/Placebo (N=5)
Toxic shock syndrome streptococcal (Infections and infestations) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBT009/Placebo (N=5)
Ecchymosis (Blood and lymphatic system disorders) | 1 (1)
Oropharyngeal pain (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Flank pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Vaginitis bacterial (Reproductive system and breast disorders) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was discontinued early due to difficulty in identifying and enrolling eligible subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No